CLINICAL TRIAL: NCT06805383
Title: Follow-up to Mailed FIT Kits
Brief Title: Randomized Trial of Follow-up to Mailed FIT Kits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Mireille Jacobson, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCHS-QIP-FOLLOWUP-FIT-KIT
Record Dates: First submitted 2025-01-13; First posted 2025-02-03 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Screening
Keywords: fecal immunochemical tests (FIT); cancer screening; Nurse follow-up

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIT Kit Only (Active Comparator): Patients sent a second FIT Kit.
  Interventions: Other: Mailed FIT Kit
- FIT Kit + Phone Call (Experimental): Patients sent a second FIT Kit and follow-up call to encourage completion and return of kit.
  Interventions: Behavioral: Phone call; Other: Mailed FIT Kit

INTERVENTIONS:
Behavioral: Phone call — Phone call to patients randomized to experimental arm.
  Arms: FIT Kit + Phone Call
Other: Mailed FIT Kit — FIT Kit mailed to patient address in EMR.

SUMMARY:
This study aims to assess whether follow-up calls can increase the return rate of mailed FIT Kits. To assess this, a randomly selected half of eligible patients were randomized to receive a follow-up call reminding the patient to return the FIT Kit.

DETAILED DESCRIPTION:
This study aims to assess whether follow-up calls can increase the return rate of mailed FIT Kits. Patients ages 45 to 59 due for colorectal cancer screening, who had not received a FIT Kit in the previous 3 months but had completed one sometime in the past and had an assigned primary care provider, were sent a FIT Kit in October of 2024. Half of patients were randomized to receive a follow-up call reminding the patient to return the FIT Kit. This work analyzes the return rate of the mailed FIT Kit, with or without phone call follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-59
* Due for colorectal cancer screening
* Not sent a FIT Kit in the past 3-months
* Previously returned a FIT Kit.

Exclusion Criteria:

* Under age 45 or over age 59;
* incarcerated;
* not due for colorectal cancer screening
* sent a FIT Kit in the past 3-months

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2135 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Return Rate | 60 Days
  FIT Kit returned to health system for processing.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Contra Costa Health Services, Martinez, California
  - Contra Costa Health, Martinez, California

IPD SHARING:
Plan to Share IPD: No
Researchers can apply for permission to use anonymized data from CCHS.